CLINICAL TRIAL: NCT03984045
Title: Sphenopalatine Ganglion Block for Treating Acute Frontal Migraine Headache in Pediatric Patients
Brief Title: SPG Block for Acute Pediatric Migraine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newark Beth Israel Medical Center (Other)
Responsible Party: Principal Investigator, Adam B Sivitz, MD, Medical Director Pediatric Emergency Medicine, Newark Beth Israel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018.42
Record Dates: First submitted 2019-06-06; First posted 2019-06-12 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Migraine in Children; Sphenopalatine Neuralgia; Migraine in Adolescence
MeSH Terms: conditions — Facial Neuralgia | interventions — Lidocaine; Prochlorperazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacy sends down drug and placebo in study preparations for administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SPG block (Experimental): SPG block performed by using qtip applicator soaked in 2% lidocaine and placed posteriorly into nasal cavity where it dwells for up to 30 min
  Interventions: Drug: Lidocaine topical
- Control (Active Comparator): Delivered through IV access obtained in all patients.
  Interventions: Drug: Prochlorperazine Injection

INTERVENTIONS:
Drug: Lidocaine topical — Intranasal 2% lidocaine delivered directly to SPG
  Arms: SPG block
Drug: Prochlorperazine Injection — intravenous prochlorperazine at 0.15mg/kg max 10 mg
  Arms: Control

SUMMARY:
This is a randomized double blind trial comparing an intranasal sphenopalatine block with 2% lidocaine to intravenous (0.15 mg/kg, max 10mg) prochlorperazine in patients greater than 10 years of age presenting to a pediatric emergency department with an acute frontal migraine headache.

DETAILED DESCRIPTION:
This is a randomized double blind trial comparing an intranasal sphenopalatine block with 2% lidocaine to intravenous (0.15 mg/kg, max 10mg) prochlorperazine in patients greater than 10 years of age presenting to a pediatric emergency department with an acute frontal migraine headache. Excluded populations include those with sickle cell, concern for CNS infection

ELIGIBILITY:
Inclusion Criteria:

- Frontal migraine headache

Exclusion Criteria:

* Non-english speaking
* Known pregnancy
* Sickle cell hemaglobinopathy
* Concern for CNS infection
* Acute febrile illness
* non-frontal headaches
* Concern for increased intracranial pressure

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to headache resolution | treatment start to patient reported resolution, up to 6 hours
  Time to headache resolution in emergency department
ED Length of stay | Registration to discharge up to 6 hours
  treatment to discharge

SECONDARY OUTCOMES:
Patient satisfaction: Rated on a Likert 100 millimeter scale | Within 6 hours from ED registration
  Patient satisfaction as determined by whether they would absolutely want treatment again (score=100), or would absolutely prefer another method (score = 0), or something in between (any mark along the 100 millimeter line)
24 hr follow up | 1 day
  Presence of headache at 24 hrs
Number of participants with treatment induced side effects | 1 day
  Recording appearance of any side effects in ED or within 24 hr follow up, such as nausea, vomiting, neck stiffness, seizure, or prolonged (greater than 6hrs) numbness.
Determine adequacy of blinding | Asked at time of patient discharge from the emergency department or at 1 hr.
  Determine whether treating physicians or patients can guess treatment arm (IN or IV arm) by simply asking the blinded patient and clinician which method they think the patient underwent. Measured by guessing one or the other arm.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Sivitz, MD, Principal Investigator — Newark Beth Israel Medical Center
Locations (1):
- Newark Beth Israel Medical Center, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No